CLINICAL TRIAL: NCT01396876
Title: Evaluation of the Effect of Hospital Clown's Performance in the Procedure Room of a Pediatric Emergency Department: A Randomized Controlled Trial
Brief Title: The Effects of Medical Clowns in Children Undergoing Blood Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-11-SR-525-CTIL
Record Dates: First submitted 2011-07-17; First posted 2011-07-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Pain; Anxiety
Keywords: Medical clown; Pediatric emergency medicine; Emergency procedures
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clown (Active Comparator): A clown is present during venipuncture
  Interventions: Behavioral: clown
- No clown (No Intervention)

INTERVENTIONS:
Behavioral: clown — a distraction technique is performed by a clown during venipuncture
  Arms: Clown

SUMMARY:
The investigators hypothesized that the participation of therapeutic clowns in the pediatric emergency department procedure room would reduce anxiety, improve the level of cooperation children can provide and avoid some of the adverse effects.

DETAILED DESCRIPTION:
Research has demonstrated that cognitive psychological techniques, including distraction, can increase pain tolerance. Humor can be an important intervention, able to reduce stress to both the child and the parent. In the last decade there has been a rapid growth in the presence of therapeutic clowns in hospital, particularly in pediatric settings. If therapeutic clowns are shown to positively affect any of the parameters being measured in this study, they should be included as aprt of the standard of care in the pediatric emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* Children needing venous blood sampling or the insertion of an intravenous canula

Exclusion Criteria:

* Children whose blood work or intravenous line must be accomplished rapidly for therapeutic reasons
* Absence of a parent during the procedure
* Abnormal development according to parents

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain score | at the end of the procedure
  recorded by the child

SECONDARY OUTCOMES:
Parental anxiety level | at the end of the procedure
  recorded by the parent
Procedure's success rate | at the end of the procedure
  recorded by the nurse
Overall report of procedure's comfort | at the end of the procedure
  recorded by the nurse

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Rimon, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel